CLINICAL TRIAL: NCT01747044
Title: Prospective Study of the Influence of the Diffuse Noxious Inhibitory Controls of the Pain on the Efficacy of Milnacipran in Fibromyalgia Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Dr. Gisèle PICKERING (MCU, PH) Center of clinical pharmacology/CIC Inserm-501 - Main investigator (Unknown); Dr Pascale PICARD/ Dr Noémie Delage / Dr Fabienne RIAUX - Center of evaluation and treatment of the pain - Investigator (Unknown); Dr Gilles DUCHEIX/ Center of clinical pharmacology/CIC Inserm-501 - Investigator (Unknown); Dr Christian DUALE/ Center of clinical pharmacology/CIC Inserm-501 - Investigator (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0130
Record Dates: First submitted 2012-11-27; First posted 2012-12-11 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Fibromylagia
Keywords: Fibromyalgia; Diffuse Noxious Inhibitory Controls; Milnacipran
MeSH Terms: conditions — Fibromyalgia | interventions — Milnacipran

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Milnacipran (Active Comparator): Milnacipran is an antidepressant known and used in major depressive disorder according to its marketing authorization but is also part of the molecules used in the treatment of chronic neuropathic pain and fibromyalgia according to the recommendations of the EULAR
  Interventions: Drug: Milnacipran
- Capsules of lactose (Placebo Comparator): placebo over a period of 8 weeks to 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Milnacipran — 100mg/day
  Arms: Milnacipran
Drug: Placebo
  Arms: Capsules of lactose

SUMMARY:
Fibromyalgia affects 0.7 to 3.3% of the adult population and 7-10 times more women than men. In France, the prevalence is 1.6% according to a French study conducted in 2009 and published in 2011 by Serge Perrot et al.

The definition of fibromyalgia was recently amended with particular consideration of cognitive and somatic symptoms, factors not involved in the initial criteria of the ACR classification. Several factors are in favor of a malfunction of the central modulation of pain and poorer performance noxious inhibitory controls descendants (DNIC: diffuse noxious inhibitory controls) have been demonstrated. In fibromyalgia patients, the DNIC (diffuse noxious inhibitory controls) are altered with less pain inhibition than controls. Dysfunction of the central pain modulation is widely described in the literature and contributes to pain complained of fibromyalgia.

According to the Recommendations of the European League Against Rheumatism (EULAR) 2006, antidepressants have a genuine analgesic efficacy in controlled studies. Milnacipran is an antidepressant known and used in major depressive disorder according to its marketing authorization but is also part of the molecules used in the treatment of chronic neuropathic pain and fibromyalgia according to the recommendations of the EULAR. A review included five double-blind studies on 4,000 participants who took 100 mg or 200 mg milnacipran or placebo over a period of 8 weeks to 24 weeks. A moderate response was obtained for 40% of participants treated for each dose of milnacipran on the criteria of "at least 30% pain relief" Impression and global change. Substantial improvement with milnacipran compared to placebo has been shown.

To date, the link between the weakening of DNIC in fibromyalgia and effectiveness of drug treatment has not been shown.

This study aims to assess the degree of impairment of DNIC in fibromyalgia patients may be predictive of the efficacy of milnacipran.

DETAILED DESCRIPTION:
Visit 1 Inclusion of the patient, Clinical examination, Evaluation of pain, basal Pain and cognitive tests

Visit 2 (can be coupled with Visit 1 if necessary) Randomisation of the patient and allocation of the treatment for 1 month.

Phone contact Visit 2 +7 days, + 15 days, +21 days Follow-up of the compliance of the treatment and collection of adverse events.

Visit 3 (follow up at 1 month) Evaluation of pain, Pain and cognitive tests End of study

ELIGIBILITY:
Inclusion Criteria:

* Patient of more than 18 years old,
* Patient with fibromyalgia

Exclusion Criteria:

* Patient with a contraindication to the administration of the milnacipran,
* Patient with a concomitant spontaneous pain not attributable of fibromyalgia,
* Patient with medical and/or surgical histories judged by the investigator not compatible with the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Pain scores on the verbal numeric scale | at T0 and T0+1 month

SECONDARY OUTCOMES:
sensitivity and pain thresholds to a mechanical stimulus | at T0 and T0+1 month
sensitivity and pain thresholds to a thermal stimulus | at T0 and T0+1 month
scores on cognitive tests | at T0 and T0+1 month
Adverse events record | at T0 and T0+1 month

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Macian N, Pereira B, Shinjo C, Dubray C, Pickering G. Fibromyalgia, milnacipran and experimental pain modulation: study protocol for a double blind randomized controlled trial. Trials. 2015 Apr 3;16:134. doi: 10.1186/s13063-015-0659-4. PMID 25873248